CLINICAL TRIAL: NCT00795886
Title: CHP-753, Rapamycin for Immunosuppression and B Cell Modulation Post Stem Cell Transplant for Acute Lymphoblastic Leukemia (ALL)
Brief Title: Rapamycin for Immunosuppression and B Cell Modulation Post Stem Cell Transplant for Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI14044
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; Cancer; Stem Cell Transplant
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental)
  Interventions: Drug: RAPAMYCIN

INTERVENTIONS:
Drug: RAPAMYCIN — Rapamycin (RAPA, RapamuneR) (sirolimus) is an immunosuppressive agent that was approved by the FDA in 1999. It is a macrocyclic lactone that is structurally similar to Tacrolimus (FK506) and binds to the same intracellular protein as FK506, FKBP1,2,3, but it has an entirely different mechanism of action and a different principal target protein. The target of the RAPA: FKBP complex is the mammalian target of rapamycin (mTOR). Unlike the calcineurin inhibitors cyclosporine (CSA) and - FK506, RAPA exerts its effects by inhibiting growth factor-driven transduction signals in the T-cell response to alloantigen, thus preventing proliferation among T and B lymphocytes3,4.
  Other Names: (RAPA, RapamuneR) (sirolimus)

SUMMARY:
Objectives:

Primary objective: Evaluate toxicity of rapamycin when used for post-bone marrow transplant graft vs. host disease prophylaxis in children with acute lymphoblastic leukemia (ALL).

Investigator initiated; four participating institutions; Phase II pilot study

DETAILED DESCRIPTION:
Objectives:

Primary objective: Evaluate toxicity of rapamycin when used for post-bone marrow transplant graft vs. host disease prophylaxis in children with acute lymphoblastic leukemia (ALL).

Rapamycin Rapamycin (RAPA, RapamuneR) (sirolimus) is an immunosuppressive agent that was approved by the FDA in 1999. It is a macrocyclic lactone that is structurally similar to Tacrolimus (FK506) and binds to the same intracellular protein as FK506, FKBP1,2,3, but it has an entirely different mechanism of action and a different principal target protein. The target of the RAPA: FKBP complex is the mammalian target of rapamycin (mTOR). Unlike the calcineurin inhibitors cyclosporine (CSA) and - FK506, RAPA exerts its effects by inhibiting growth factor-driven transduction signals in the T-cell response to alloantigen, thus preventing proliferation among T and B lymphocytes3,4. This action is at a later stage in T cell mediated response than that of CSA or FK506. Important cyclin-dependent signaling kinases are blocked, which results in cell cycle arrest between G1 and S phase. RAPA prevents factor dependent growth of activated T cells, but does not prevent the autocrine production or release of growth factors from activated T cells. Rapamycin has been studied in clinical trials of solid organ allografts, and have been shown to prolong allograft survival by inhibiting host CD4+ and CD8+ T cell expansion5, 6. RAPA has synergistic immunosuppressive properties when used with CSA or FK506, and its use allows lower doses of the more nephrotoxic calcineurin inhibitors to accomplish decreased rejection. The use of full dose calcineurin inhibitors with RAPA can result in nephrotoxicity, but these agents can be safely used at a reduced dose with RAPA.

Our goal with Rapamycin is to achieve two necessary ends with one medication: a leukemic precursor effect (see above), and prevention of graft vs. host disease (GVHD). With CSA OR FK506, acute GVHD develops in approximately 40% of pediatric matched related donor recipients, and the majority is mild and easily controllable by the addition of methylprednisolone or prednisone. At Children's hospital of Philadelphia (CHOP), "short course" methotrexate in addition to CSA OR FK506 is given only to patients >14 years, or those with older donors. Chronic GVHD occurs in approximately 20% of pediatric matched related donor recipients, and 75% of this is limited to skin. Therefore, the use of RAPA in this group may accomplish adequate immunosuppression so as to prevent GVHD, as well as provide anti- B and anti-T cell malignancy effect. RAPA may also prove less toxic than the calcineurin inhibitors as well, in which both nephrotoxicity and neurotoxicity remain serious side effects.

Allogeneic bone marrow transplantation for children with ALL Children who have very high-risk features, such as t(4;11) or t(9;22), or those who relapse while on chemotherapy are rarely cured by chemotherapy alone. These patients, as well as those beyond second remission, are generally referred for allogeneic stem cell transplantation. Approximately 25-30% of these patients will have a matched sibling donor. Matched sibling, matched unrelated, and cord blood donor bone marrow transplant results in approximately 40-60% of patients surviving disease free, but relapse remains the largest obstacle to cure. Rapamycin, with its apoptotic effects upon B cell precursor malignancies, may prove effective in decreasing the incidence of relapse in these patients, particularly when used in a state of minimal residual disease post transplant. We expect to treat approximately 10 patients with ALL yearly with matched related donor BMT between the four centers involved in this study.

Rapamycin studies in conjunction with a calcineurin inhibitor (CSA or FK506) At the Dana Farber Cancer Institute (DFCI), 50 patients with related, human leukocyte antigen (HLA) matched peripheral stem cell transplants were studied using the combination of FK506 and repaying. The hypothesis tested was that the omission of methotrexate would not increase the rate of GVHD, and would reduce toxicity. The rate of grade II-IV acute GVHD was 16%, and III-IV 5%, which is extremely favorable for adults. Transplant related mortality at 100 days was 5%.

This study was done following an earlier study of low dose methotrexate in the higher risk unrelated donor transplant patient. This study showed that rapamycin provided excellent GVHD prevention in the high-risk cohort.

We will substitute FK506 for cyclosporine as per the Boston experience. This will be considered a standard practice within our division to increase patient compliance and comfort. This does not increase risk to patients, as oral FK506 is better tolerated RAPA and FK506 appear to be synergistic which may result in better GVHD prophylaxis.

Study Procedures:

Conditioning:

1. Thiotepa 5 mg/kg days -7, -6. Given IV over 4 hours. Cyclophosphamide 60 mg/kg days -5, -4. Given over 1 hour IV with routine supportive care.
2. Total body irradiation (TBI) 200 cGy/fraction x 6 fractions given over 3 days*. Testicular boost 400 cGy may be given for males. Patients with prior CNS disease and no prior central nervous system (CNS) irradiation: 600 cGy prior to starting conditioning. *TBI may be given before or after Thiotepa and cyclophosphamide. If given before Stem cells are to be given 48 hours after the end of cyclosphosphamide.

Graft vs. Host Disease Prophylaxis:

1. Tacrolimus IV by continuous infusion .03mg/kg per day beginning day -3. Target serum levels between 5-10 patients will switch to oral form when tolerating PO's ("Per Os" or "By mouth".
2. Methotrexate 5mg/m2 will be given IV on days 1, 3, and 6 for all patients and on day 11 for patients receiving unrelated donor marrow.
3. Rapamycin day 0 with dosing as follows: 2.5 mg/m2/d (4mg/d max) PO daily.

Absent GVHD Immune Suppression Weaning:

1. Tacrolimus: Matched sibling donor allograft taper at day +42 over 6-8wks. Mismatched or unrelated allograft or cord blood taper at day +100 to be off by day +180.
2. Sirolimus: At day + 180 wean over 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients' ages (0 - 21 years) with lymphoid malignancies considered for allogeneic bone marrow transplant from HLA-identical sibling donor, single antigen mismatched related or unrelated donor marrow /peripheral blood stem cell (PBSC) or cord blood available for marrow donation.

   First remission:
   * if remission not achieved by day28
   * high risk cytogenetic features, including t(9;22) or t(4;11) Second or third remission
2. Signed informed consent.

Exclusion Criteria:

1. Organ criteria:

1. Cardiac: ECHO shortening fraction <27%
2. Renal: Creatinine clearance <60 ml/min/1.73 m2
3. Hepatic: Bilirubin >1.5 mg/dl, transaminases <3x normal
4. Infection: active viral, fungal or bacterial infection including HIV.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2005-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pulsipher, MD, Principal Investigator — Primary Children's Hospital
Locations (1):
- Primary Children's Medical Center, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between Aug 2003 and Aug 2008 from 4 pediatric centers in the United States. (Childrens Hospital of Philadelphia; Methodist Childrens Hospital of South Texas (San Antonio); Primary Childrens Medical Center (Salt Lake City); and Childrens Hospital of Pittsburgh.
Groups:
- Rapamycin: This includes all study participants.
Period: Overall Study
Arm/Group | Rapamycin
Started | 63
Completed | 53
Not Completed | 10
Not completed — Death | 10

BASELINE CHARACTERISTICS:
Arm/Group | Rapamycin
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 61
  Between 18 and 65 years | 2
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.9 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Transplant-related Mortality
Description: Death not associated with relapse. We determined that if transplant related mortality(TRM) 25% at day 100 or if Grade III-IV (severe, life threatening, or disabling) acute GVHD was >30% a stopping rule would be triggered.
Time Frame: 24 months after transplant
Population: All participants enrolled in the trial.
Measure: Number; unit: participants
Groups:
- Rate of Transplant Related Mortality: All participants enrolled in the trial
Arm/Group | Rate of Transplant Related Mortality
Number analyzed (Participants) | 63
participants | 8

2. Secondary Outcome: Percentage of Patients Developing Acute Graft vs. Host Disease (GVHD)
Description: Cumulative incidence of Grade 2-4 acute GVHD at 180 days.
Time Frame: 180 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rapamycin
Number analyzed (Participants) | 63
percentage of participants | 38 [26 to 50]

3. Primary Outcome: Two Year Overall Survival
Description: The probability that a given patient will be alive two years after transplantation. The Kaplan-Meier product limit method was used to compute the probability of overall survival to 2 years. Greenwood's formula was used to compute the standard error.
Time Frame: 24 months after transplant
Population: All patients enrolled in study.
Measure: Mean (Standard Error); unit: probability
Arm/Group | Rapamycin
Number analyzed (Participants) | 63
probability | 0.73 (0.058)

ADVERSE EVENTS:
Time Frame: Over the 3 years of the trial and two years after completing.
Arm/Group | Rapamycin
Serious Adverse Events (participants affected / at risk) | 8/63
Other Adverse Events (participants affected / at risk) | 3/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapamycin (N=63)
Transplant related mortality (Blood and lymphatic system disorders) | 8 (8) — Death not related to relapse
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapamycin (N=63)
Venoocclusive Disease (Hepatobiliary disorders) | 3 (3) — Looking at non-severe VOD. Important to understand this as it has been noted in a portion of patients using sirolimus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No